CLINICAL TRIAL: NCT05038735
Title: EPIK-B5: A Phase III, Randomized, Double-blind, Placebo-controlled Study of Alpelisib in Combination With Fulvestrant for Men and Postmenopausal Women With HR-positive, HER2-negative Advanced Breast Cancer With a PIK3CA Mutation, Who Progressed on or After Aromatase Inhibitor and a CDK4/6 Inhibitor
Brief Title: Study to Assess the Efficacy and Safety of Alpelisib Plus Fulvestrant in Participants With HR-positive (HR+), HER2-negative, Advanced Breast Cancer After Treatment With a CDK4/6 Inhibitor and an Aromatase Inhibitor.
Acronym: EPIK-B5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CBYL719C2303; 2023-509133-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Alpelisib; Fulvestrant; Advanced breast cancer; Phase III; HR-positive; HER-2 negative; CDK4/6 inhibitor; PIK3CA mutation; Progression free survival; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpelisib plus fulvestrant (Experimental): Alpelisib 300 mg orally once daily on a continuous dosing schedule, in a 28-day cycle + fulvestrant 500 mg as intramuscular injection on Cycle 1 Day 1 and 15, and on Day 1 on every Cycle thereafter, in a 28 days cycle.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant
- Alpelisib-matching placebo plus fulvestrant (Placebo Comparator): Alpelisib-matching placebo orally once daily on a continuous dosing schedule, in a 28-day cycle + fulvestrant 500 mg as intramuscular injection on Cycle 1 Day 1 and 15 and on Day 1 on every Cycle thereafter, in a 28 days cycle.
  After Protocol Amendment 5 is implemented, alpelisib matching-placebo will no longer be supplied or administered once participants have been unblinded.
  Interventions: Drug: Fulvestrant; Drug: Alpelisib-matching placebo

INTERVENTIONS:
Drug: Alpelisib — Alpelisib (tablets) administered at 300mg orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 day cycle.
  Arms: Alpelisib plus fulvestrant
Drug: Fulvestrant — Fulvestrant (prefilled syringe) 500mg administered intramuscularly at Cycle 1 Day 1 and 15 and then at Day 1 of each subsequent cycle (each cycle is 28 days).
Drug: Alpelisib-matching placebo — Alpelisib-matching placebo (tablets) administered orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 day cycle.
  After Protocol Amendment 5 is implemented, alpelisib matching-placebo will no longer be supplied or administered once participants have been unblinded.
  Arms: Alpelisib-matching placebo plus fulvestrant

SUMMARY:
The purpose of this study is to complement Study CBYL719C2301 (SOLAR-1) and obtain more comprehensive data on the efficacy and safety of alpelisib (BYL719) in combination with fulvestrant compared with placebo plus fulvestrant in men or postmenopausal women with HR-positive, HER2-negative advanced breast cancer with a PIK3CA mutation who progressed or relapsed on or after treatment with an AI plus a CDK4/6 inhibitor.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, international, multi-center trial. Men and postmenopausal women will be randomized to either alpelisib plus fulvestrant or alpelisib-matching placebo plus fulvestrant. Randomization will follow a 1:1 randomization ratio and be stratified by presence of lung and/or liver metastases (yes vs. no) and setting at last prior CDK4/6 inhibitor therapy (adjuvant vs metastatic).

Study treatment with alpelisib plus fulvestrant or alpelisib-matching placebo plus fulvestrant will be initiated on Cycle 1 Day 1, and will continue until disease progression per RECIST v1.1 as per BIRC assessment, start of new antineoplastic therapy, death, lost to follow-up, or withdrawal of consent. A cycle is defined as 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is an adult ≥ 18 years old at the time of informed consent and has signed informed consent before any trial related activities and according to local guidelines.
* Participant has a histologically and/or cytologically confirmed diagnosis of ER+ and/or PgR+ breast cancer by local laboratory.
* Participant has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescent in situ hybridization (FISH), Chromogenic in situ hybridization (CISH), or Silver-enhanced in situ hybridization (SISH)) test is required by local laboratory testing.
* Participant has at least one measurable lesion as per RECIST v1.1 criteria as assessed by Investigator (a lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation).
* Participant has recurrence or progression of disease during or after combined AI (i.e. letrozole, anastrozole, exemestane) and CDK4/6 inhibitor therapy. The combined AI and CDK4/6 inhibitor therapy does not need to be the latest treatment regimen (including adjuvant setting).
* Participant has received ≤ 2 prior lines of systemic therapies overall in the metastatic setting, of which a maximum of 1 line of prior treatment with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy) is permitted.
* The presence of PIK3CA mutation(s) determined in tumor tissue prior to enrollment either by a Novartis designated laboratory or in tumor tissue or plasma ctDNA by a local laboratory using a Food and Drug Administration (FDA)-approved PIK3CA Companion Diagnostics (CDx) test for alpelisib or the CE-IVD QIAGEN Therascreen® PIK3CA RGQ PCR test.
* If female, then the participant must be in postmenopausal status.

Key Exclusion Criteria:

* Participant with symptomatic visceral disease or any disease burden that makes the participant ineligible for endocrine therapy (ET) per the Investigator's best judgment.
* Participant who relapsed with documented evidence of progression more than 12 months from completion of (neo)adjuvant endocrine/endocrine-based therapy with no treatment for metastatic disease.
* Participant has received prior treatment with fulvestrant, any oral selective estrogen receptor degrader (SERD), any Phosphatidylinositol-3-Kinase (PI3K), mammalian Target of Rapamycin (mTOR) or Protein Kinase B (AKT) inhibitor.

Other Inclusion and Exclusion Criteria do apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on BIRC assessments and using RECIST v1.1 criteria | From randomization to date of the first documented progression or death due to any cause, assessed up to a maximum duration of 60 months.
  Progression-free survival (PFS) is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS will be assessed by the Blinded Independent Review Committee (BIRC) according to RECIST 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death up to a maximum duration of 60 months
  Overall survival (OS) is defined as the time from randomization to the date of death due to any cause
Overall response rate (ORR) with confirmed response based on BIRC assessments and using RECIST v1.1 criteria | From the date of randomization up to a maximum duration of 60 months
  Overall response rate (ORR) with confirmed response is defined as the proportion of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), as per BIRC and according to RECIST 1.1
Clinical benefit rate (CBR) with confirmed response based on BIRC assessments and using RECIST v1.1 criteria | From the date of randomization up to a maximum duration of 60 months
  Clinical benefit rate (CBR) with confirmed response is defined as the proportion of participants with a best overall response of confirmed CR or PR, or SD lasting for a duration of at least 24 weeks. CR, PR and SD are defined as per BIRC review according to RECIST 1.1
Duration of response (DOR) with confirmed response based on BIRC assessments and using RECIST v1.1 criteria | From first documented response to the date of first progression or deaths, up to a maximum duration of 60 months
  Duration of response (DOR) with confirmed response only applies to participants whose best overall response is confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1 based on tumor response data per BIRC review. The start date is the date of first documented response of CR or PR and the end date is defined as the date of the first documented progression or death due to underlying cancer.
Time to response (TTR) based on BIRC assessments and using RECIST v1.1 criteria | From the date of randomization to the first documented response up to a maximum duration of 60 months
  Time to response (TTR) is defined as the time from the date of randomization to the first documented response of either complete response (CR) or partial response (PR), which must be subsequently confirmed. CR and PR are based on tumor response data as per BIRC review and according to RECIST 1.1
PFS based on BIRC assessment and using RECIST v1.1 criteria for participants by PIK3CA mutation status | From the date of randomization up to a maximum duration of 60 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS will be assessed by the Blinded Independent Review Committee (BIRC) according to RECIST 1.1. Results will be presented by PIK3CA mutation status measured in circulating tumor deoxyribonucleic acid (ctDNA) collected at baseline.
Time to definitive deterioration of Eastern Cooperative Oncology Group (ECOG) performance status (PS) from baseline | From the date of randomization up to maximum duration of 60 months
  Time to definitive deterioration of Eastern Cooperative Oncology Group (ECOG) performance status (PS) from baseline is defined as the time from the date of randomization to the date when ECOG PS has definitively worsened by at least one category compared to baseline. Deterioration is considered definitive if there is no subsequent improvement in ECOG PS back to the baseline category or better.
Time to definitive (10%) deterioration in the global health status/Quality of Life (QoL) and symptom scale scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30) | From the date of randomization up to maximum duration of 60 months
  Time to definitive (10%) deterioration in global health status/Quality of Life (QoL) and symptom scale scores of the EORTC QLQ-C30 is defined as the time from the date of randomization to the date of the first occurrence of at least a 10% worsening from baseline in the global health status/QoL or symptom scale scores, with no subsequent improvement above this threshold during treatment or until death from any cause. The EORTC QLQ-C30 is a validated questionnaire assessing cancer patients' quality of life over the past week, comprising 30 items across 5 functional scales, 3 symptom scales, 6 single items, and a global health status/QoL scale. Scores range from 0 to 100, with higher scores indicating a higher response level.
Change from baseline in global health status/QoL and symptom scale scores of the EORTC QLQ-C30 | From the date of randomization up to maximum duration of 60 months
  Change from baseline in global health status/Quality of Life (QoL) and symptom scale scores of the EORTC QLQ-C30 refers to the variation in scores from baseline across domain scores, health states, overall health status, and index values at each assessment timepoint. The EORTC QLQ-C30 is a validated questionnaire designed to assess the quality of life of cancer patients over the past week. It includes 30 items comprising 5 functional scales, 3 symptom scales, 6 single items, and a global health status/QoL scale. Each scale and item is scored from 0 to 100, with higher scores indicating a higher response level.
Time from randomization to objective tumour progression on next line treatment or death from any cause (PFS2) | From the date of randomization up to maximum duration of 60 months
  Time from randomization to objective tumor progression on next-line treatment or death from any cause (PFS2) is defined as the time from the date of randomization to the earliest occurrence of either documented disease progression on next-line therapy, as assessed by the investigator, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- Belgium (5):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Ottawa, Ontario
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Aalborg, Denmark
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
- France (8):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Valenciennes
- Germany (5):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Lübeck
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Dublin, Ireland
- Italy (13):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Bydgoszcz, Poland
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Floreşti, Cluj, Romania
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Spain (8):
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com